CLINICAL TRIAL: NCT00000720
Title: A Double-Blind, Placebo-Controlled Trial To Evaluate Intravenous Gamma Globulin in Children With Symptomatic HIV Infection Receiving Zidovudine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 051; 11025 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Placebos; Infusions, Intravenous; Gamma-Globulins; Combined Modality Therapy; Acquired Immunodeficiency Syndrome; Zidovudine; Bacterial Infections; Immunization, Passive
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Bacterial Infections | interventions — Immunoglobulins; Zidovudine

INTERVENTIONS:
Drug: Globulin, Immune
Drug: Zidovudine

SUMMARY:
To evaluate the clinical, immunologic, and virologic effects of oral zidovudine (AZT) plus intravenous immunoglobulin (IVIG) versus AZT plus placebo (albumin). It is estimated that by 1991, there may be 10,000 to 20,000 HIV-infected children in the United States. HIV infection in children is most often associated with symptomatic disease and poor prognosis. Treatment with antiviral therapy may be effective in changing the course of disease and decreasing mortality in this vulnerable population. AZT treatment has been shown to decrease mortality and the frequency of opportunistic infections in certain adult AIDS patients; therefore, it is likely that children may also benefit from this antiviral therapy. In addition, bacterial infections are frequently found in HIV-infected children. Because pooled human serum immunoglobulin, another name for antibodies, is effective in reducing bacterial infection in patients with defects of immunity, it may reduce the rate of bacterial infection in HIV-infected children as well. In this study, AZT will be administered together with IVIG to determine safety, tolerance, and efficacy of the combined treatment.

DETAILED DESCRIPTION:
It is estimated that by 1991, there may be 10,000 to 20,000 HIV-infected children in the United States. HIV infection in children is most often associated with symptomatic disease and poor prognosis. Treatment with antiviral therapy may be effective in changing the course of disease and decreasing mortality in this vulnerable population. AZT treatment has been shown to decrease mortality and the frequency of opportunistic infections in certain adult AIDS patients; therefore, it is likely that children may also benefit from this antiviral therapy. In addition, bacterial infections are frequently found in HIV-infected children. Because pooled human serum immunoglobulin, another name for antibodies, is effective in reducing bacterial infection in patients with defects of immunity, it may reduce the rate of bacterial infection in HIV-infected children as well. In this study, AZT will be administered together with IVIG to determine safety, tolerance, and efficacy of the combined treatment.

The study includes 250 children, 3 months to 12 years of age. All participants receive oral AZT. IVIG or intravenous placebo is administered every 28 days. Patients are followed for the development of serious bacterial infection, as well as for a number of factors relating to safety, tolerance, progression of disease, and survival. This is an outpatient study conducted over a minimum 100-week period. The children are evaluated every 2 weeks for the first 8 weeks, and monthly thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Benadryl and/or acetaminophen may be given before and during intravenous immunoglobulin (IVIG) infusion in patients demonstrating mild reactions during infusion.
* Acetaminophen for short-term fever and pain.
* Zidovudine (AZT).
* Steroids.
* Oral or systemic (swish and swallow) nystatin.
* Maintenance therapy for fungal disease or tuberculosis.
* Prophylaxis for a previous episode of Pneumocystis carinii pneumonia (PCP) including the use of trimethoprim / sulfamethoxazole (TMP / SMX). The dosage is specified as TMP 75 mg/m2 twice daily 3 times a week and SMX 375 mg/m2 twice daily 3 times a week.
* Recommended:
* Children with AIDS and / or CD4 count = or < 500 cells/mm3 should receive primary PCP prophylaxis as described.

Concurrent Treatment:

Allowed:

* Blood transfusion for hemoglobin < 8 g/dl and hematocrit < 24 percent or bone marrow suppression.
* Supplemental oxygen with a prestudy PaO2 < 70 mmHg.

Children must have one or more of the indicator diseases of AIDS; however, there must be an absence of acute opportunistic infection and an absence of bacterial infection requiring treatment at the time of entry into the study.

* Children with lymphoid interstitial proliferation (LIP) are excluded from enrollment unless they have had additional AIDS-defining opportunistic infections, meet ARC criteria, have had two or more serious bacterial infections in the 12 months prior to study entry, have evidence of HIV encephalopathy, or are currently on supplemental oxygen and steroids with a pre-treatment PaO2 < 70 mm Hg.
* Children with concurrent LIP and ARC are eligible for inclusion. Thrombocytopenia is an exclusion except if it is HIV-associated.
* Children randomized prior to their 13th birthday are eligible.
* All lab values must be within 4 weeks of study entry.

Prior Medication:

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following will be excluded:

* Lymphoid interstitial proliferation (LIP) not requiring steroids and supplemental oxygen or with other lymphoproliferative diseases as their sole clinical evidence of HIV infection.
* Known hypersensitivity to immunoglobulin.
* Active HIV thrombocytopenia requiring IVIG therapy.

Concurrent Medication:

Excluded:

* Chronic acetaminophen.
* Drugs that are metabolized by hepatic glucuronidation should not be used for more than 24 hours without notifying the study physician.
* Antibacterial prophylaxis for otitis, sinusitis, or urinary tract infection.
* Prophylaxis treatment for Pneumocystis carinii pneumonia (PCP) prior to the first episode of laboratory-documented PCP.
* Immunoglobulin (IVIG) therapy required for active HIV thrombocytopenia.

Patients with the following will be excluded:

* Lymphoid interstitial proliferation (LIP) not requiring steroids and supplemental oxygen or with other lymphoproliferative diseases as their sole clinical evidence of HIV infection.
* Known hypersensitivity to immunoglobulin.
* Active HIV thrombocytopenia requiring IVIG therapy.
* Inability to establish or maintain intravenous access.
* Lack of parental or guardian authorization for intravenous access.

Prior Medication:

Excluded within 4 weeks of study entry:

* Any other experimental therapy.
* Other antiretroviral agents.
* Drugs which cause prolonged neutropenia or significant nephrotoxicity.
* Immunoglobulins.
* Immunomodulating agents.

Active alcohol or drug abuse.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250
Dates: Study Completion 1993-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spector, SA, Study Chair
Locations (51):
- United States (48):
  - Kaiser Permanente / UCLA Med Ctr, Downey, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - Martin Luther King Jr Gen Hosp / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Stanford Univ School of Medicine, Menlo Park, California
  - Children's Hosp of Oakland, Oakland, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Northern California Pediatric AIDS Treatment Ctr / UCSF, San Francisco, California
  - Olive View Med Ctr, Sylmar, California
  - Univ of Connecticut Health Ctr / Pediatrics, Farmington, Connecticut
  - Emory Univ School of Medicine, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - SUNY / Health Sciences Ctr at Brooklyn / Pediatrics, Brooklyn, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Schneider Children's Hosp / Long Island Jewish Med Ctr, New Hyde Park, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Univ Babies' Hosp, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Lincoln Hosp Ctr / Pediatrics, The Bronx, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Westchester Hosp / New York Med College / Pediatrics, Valhalla, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of Seattle, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - San Juan City Hosp, San Juan
  - UPR Children's Hosp / San Juan City Hosp, San Juan

REFERENCES:
- [Background] Connor E, McSherry G. Treatment of HIV infection in infancy. Clin Perinatol. 1994 Mar;21(1):163-77. PMID 7912175
- [Background] Mofenson LM, Moye J Jr. Intravenous immune globulin for the prevention of infections in children with symptomatic human immunodeficiency virus infection. Pediatr Res. 1993 Jan;33(1 Suppl):S80-7; discussion S87-9. doi: 10.1203/00006450-199305001-00464. PMID 8433880
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891
- [Background] Spector SA, Gelber RD, McGrath N, Connor EM, Wara DW, Balsley JF. Results of a double-blind placebo-controlled trial to evaluate intravenous gamma globulin in children with symptomatic HIV infection receiving zidovudine (ACTG 051). The Pediatric AIDS Clinical Trials Group and the NICHD Pediatric HIV Centers. Int Conf AIDS. 1993 Jun 6-11;9(1):48 (abstract no WS-B05-6)
- [Background] Spector SA, Gelber RD, McGrath N, Wara D, Barzilai A, Abrams E, Bryson YJ, Dankner WM, Livingston RA, Connor EM. A controlled trial of intravenous immune globulin for the prevention of serious bacterial infections in children receiving zidovudine for advanced human immunodeficiency virus infection. Pediatric AIDS Clinical Trials Group. N Engl J Med. 1994 Nov 3;331(18):1181-7. doi: 10.1056/NEJM199411033311802. PMID 7935655